CLINICAL TRIAL: NCT00670150
Title: Phase II Study of NRX 195183 Induction and NRX 195183 Combined With Arsenic Trioxide (As2o3) as Initial Consolidation Therapy Followed by Continuous NRX 195183 Maintenance Therapy for Patients With Untreated Acute Promyelocytic Leukemia
Brief Title: New Retinoid Agent Combined With Arsenic Trioxide for Untreated Acute Promyelocytic Leukemia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: sponsor withdrew support
Sponsor: University of Southern California (Other)
Collaborators: Sponsor Name Pending (Industry)
Responsible Party: Dr. Dan Douer, University of Southern California
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9L-07-12
Record Dates: First submitted 2008-04-28; First posted 2008-05-01 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2015-10

CONDITIONS: Acute Promyelocytic Leukemia
MeSH Terms: conditions — Leukemia, Promyelocytic, Acute | interventions — Arsenic Trioxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: NRX 195183 (retinoid analogue) — 30mg/m2 PO daily x 3mo.in Induction, then daily with consolidation
Drug: Arsenic Trioxide — 0.15mg/kg/day over 2hrs VI on day 1-5 x 4 weeks. 2 weeks rest then repeat x 3 more cycles.

SUMMARY:
The safety and efficacy of combining NRX 195183 with arsenic trioxide in treating untreated APL will be assessed.

DETAILED DESCRIPTION:
The primary objectives of this study are in newly diagnosed APL patients:

* To evaluate the efficacy (complete and molecular response rates) and toxicity of NRX 195183 in induction therapy
* To evaluate the efficacy (molecular response rates) and toxicity of NRX 195183 in combination with arsenic trioxide (As2O3) in consolidation therapy.
* To evaluate the efficacy (event free-survival, disease-free survival) and toxicity of NRX 195183 as maintenance therapy for patients with APL who achieve a molecular complete response.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis Patients must have a clinical diagnosis of acute promyelocytic leukemia (APL) morphology or FAB M3 variant confirmed by RT-PCR assay for PML-RARα or chromosome analysis/FISH showing t(15:17) translocation. A patient may be entered prior to confirmatory studies, but a patient who is subsequently found to be PML-RARα negative will be removed from protocol treatment.
* Prior Treatment The patient must not have received any systemic definitive treatment for APL, including cytotoxic chemotherapy, retinoids or arsenic trioxide. Prior therapy with corticosteroids, hydroxyurea or leukapheresis will not exclude the patient.
* Age: Patients must be of age eighteen (18) or above.
* Other Criteria

  * Patients must have the following laboratory values:

    * Bilirubin equal or less than 1.5 times the upper limit of normal.
    * Creatinine equal or less than 1.5 times the upper limit of normal
* Pregnancy / Nursing Status

  * Patients entered into this study should be non-pregnant and non-nursing and should not plan on becoming pregnant while on treatment. Treatment under this protocol would expose an unborn child to significant risks. treatment. Women and men of reproductive potential should agree to use an effective means of birth control. There is an extremely high risk of fetal malformation if pregnancy occurs while on treatment in any amount with retinoid drugs even for short periods.

Exclusion Criteria:

* Non-APL, AML patients should be excluded from the study.
* Other serious illnesses which would limit survival to 1 year.
* Psychiatric conditions which would prevent compliance with treatment or informed consent.
* Uncontrolled or severe cardiovascular disease. This would include history of a recent acute myocardial infarction, uncontrolled congestive heart failure, or active angina.
* AIDS or HIV positive patients, although HIV test is not required for accrual.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-05; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is achieving a partial or complete response | Bone marrow biopsies will be done monthly during induction

SECONDARY OUTCOMES:
Safety and feasibility | Twice weekly during induction and then weekly during consolidation

CONTACTS AND LOCATIONS:
Overall Officials: Dan Douer, MD, Principal Investigator — University of Southern California
Locations (1):
- USC/Norris Comprehensive Cancer Center, Los Angeles, California, United States